CLINICAL TRIAL: NCT06688071
Title: FAPI PET/CT in Various FAP-Related Disease Patients
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University General Hospital
Other Study IDs: TJMUGH-01
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: FAP-related Disease; Tumor; Positron Emission Tomography; Metastasis
Keywords: PET/CT; FAP; FAPI
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Single Group Assignment — 68Ga-DOTA/NOTA-FAPI-04 Each subject receive a single intravenous injection of 68Ga/18F-FAPI, and undergo PET/CT imaging within the specificed time.

SUMMARY:
To evaluate the potential usefulness of 68Ga/18F-FAPI positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various FAP-related disease patients.

DETAILED DESCRIPTION:
Subjects with various FAP-related disease patients underwent 68Ga/18F-FAPI PET/CT either for an initial assessment or for recurrence detection. Lesions uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga/18F-FAPI PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled FAPI PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions; (ii) patients with pregnancy; (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled FAPI PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of FAPI for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of FAPI PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No